CLINICAL TRIAL: NCT05081193
Title: A Phase II Study Assessing the Safety and Efficacy of Oral Testosterone Undecanoate Followed by Enzalutamide as Therapy for Men With Metastatic Castrate Resistant Prostate Cancer
Brief Title: Safety and Efficacy of Oral Testosterone Undecanoate Followed by Enzalutamide as Therapy for Men With Metastatic Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Clarus Therapeutics, Inc. (Industry); Allegheny Health Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2178; IRB00284702 (Other: Johns Hopkins Medicine)
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Oral Testosterone Therapy; Enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone undecanoate; Testosterone Propionate; enzalutamide

STUDY DESIGN:
Intervention Model Description: Oral Testosterone Therapy-396 mg given twice per day on days 1-7 and 15-21 of a 28 day cycle until radiographic progression. After a 21 day washout period, Enzalutamide therapy given at 160 mg once daily will be taken for a maximum of 6 cycles while on study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Testosterone Therapy given until radiographic progression followed by Enzalutamide Therapy (Experimental): Oral Testosterone Therapy-396 mg given twice per day on days 1-7 and 15-21 of a 28 day cycle until radiographic progression. After a 21 day washout period, Enzalutamide therapy given at 160 mg once daily will be taken for a maximum of 6 cycles while on study.
  Interventions: Drug: Testosterone Undecanoate; Drug: Enzalutamide

INTERVENTIONS:
Drug: Testosterone Undecanoate — 198mg taken twice daily
  Other Names: Jatenzo
Drug: Enzalutamide — 160mg taken once daily
  Other Names: Xtandi

SUMMARY:
Previous studies of high dose testosterone therapy given intramuscularly to men with metastatic castrate resistant prostate cancer suggest that high serum levels of testosterone may be required for clinical response. This injection regimen was given as one dose of 400mg injection every 28 days, which initially produces high serum testosterone levels but these levels drop to a varying degree in some men over the 28-day cycle.

In this 30 patient trial will analyze the effects of oral testosterone therapy in men with metastatic castrate resistant prostate cancer taken on a schedule of seven days of oral testosterone therapy followed by seven days of no therapy for a twenty-eight day cycle. This therapy will be given for three 28 day cycles consecutively followed by radiographic scans to evaluate the metastatic disease. Patients will be allowed to continue on this therapy until the patients show signs of radiographic progression. If the patients show signs of radiographic progression after the first three cycles, the patients will stop taking the oral testosterone therapy and begin taking enzalutamide therapy. Enzalutamide therapy will be taken for three 28 day cycles, then radiographic scans will be taken. If there are no signs of radiographic progression, patients can continue to take enzalutamide therapy for an additional 3 cycles while on study. Patients with continued PSA or objective response will come off study but continue on enzalutamide as standard of care therapy.

This study will help the investigators to understand if treating these men with the highest FDA approved dose of oral testosterone therapy will achieve similar and sustained high levels of serum testosterone that will produce similar or enhanced therapeutic response to the therapy when compared to the serum testosterone levels found in the previous injection therapy trials.

DETAILED DESCRIPTION:
Metastatic prostate cancer is a highly significant disease that claims the lives of approximately 30,000 American men each year. Androgen Deprivation Therapy (ADT) is initially very effective but is never curative as all men eventually develop castrate resistant prostate cancer (CRPC). A major factor driving resistance is the ability of prostate cancer (PCa) cells to adapt to the chronic low androgen conditions by upregulating androgen receptor (AR) activity through overexpression, gene amplification and expression of truncated, transcriptionally active AR variants that lack the ligand-binding domain. Persistent signaling through AR makes CRPC sensitive to more potent inhibition of AR by abiraterone acetate or second generation anti-androgens such as enzalutamide. Yet these therapies have a limited duration of benefit prior to development of resistance, often through further increase in AR levels.

While this marked upregulation of AR can drive resistance, the investigators have demonstrated that it also creates a therapeutic vulnerability to exposure to high levels of androgen. However, the investigators have also found that sustained exposure of CRPC to supraphysiological levels of androgens results in downregulation of AR and acquired resistance to this therapy. Therefore the investigators have developed a therapy called Bipolar Androgen Therapy (BAT) in which testosteronecypionate 400 mg IM is administered every 28 days to result in cycling from supraphysiological (>1500 ng/dL) to near-castrate levels. The rationale for cycling was that high serum T would kill high AR expressing CRPC while low serum T would prevent adaptation to high T and kill low AR expressing CRPC.

To date the investigators have treated approximately 250 men with BAT across four completed studies in asymptomatic men with CRPC. The key findings have been that BAT: (a) could be safely administered; (b) did not produce symptomatic disease progression; (c) produced sustained PSA and objective responses in approximately 30-40% of patients; (d) re-sensitized and prolonged response of patients to subsequent antiandrogen therapy. While ADT for advanced PCa often produces debilitating sexual and metabolic side effects, another highly significant feature of this approach is that BAT can make men feel remarkably better by decreasing fatigue, increasing physical activity and restoring libido and sexual function. BAT also produced favorable effects on body composition by increasing skeletal muscle mass and decreasing subcutaneous and visceral fat. Thus, incorporation of BAT into the treatment paradigm has the potential to improve the quality of life and well-being of PCa patients and minimize the morbidity from the metabolic sequelae produced by androgen ablative therapies.

The studies performed to date demonstrate the safety and efficacy of high dose T in men with metastatic CRPC who are progressing on androgen ablative therapy. The investigators' limited data suggests that high serum levels of T may be required for clinical response. This high level has is achieved through intramuscular (IM) administration of testosterone cypionate at the highest FDA-approved dose of 400 mg every 28 days. This regimen initially produces high serum T levels but these levels drop to a varying degrees approaching near castrate levels in some men over a 28-day cycle. To date, the investigators have not tested whether more rapid cycling of serum T would produce similar or improved therapeutic response in this patient population. Additional issues with IM testosterone are (1) it requires patients to come to hospital every 28 days for injection, (2) has highly variable pharmacokinetics, (3) can cause physical discomfort from IM injections.

Recently two novel oral testosterone (OT) agents were developed for the treatment of male hypogonadism. Historically, an oral option for testosterone replacement therapy was unavailable because of risks of liver toxicity, including cholestasis and jaundice, associated with earlier developed 17-alpha-alkylated oral analogs. These novel oral agents feature specialized formulations that avoid adverse hepatic effects. In clinical trials, both oral agents produced no significant adverse effects on liver function tests. The investigators have formed a collaborative partnership with Clarus Therapeutics, the makers of Jatenzo, an oral lipoprotein-coated testosterone undecanoate (OT) formulation that was FDA-approved in December 2019 as T-replacement therapy. Published pharmacokinetic data demonstrate that OT can produce supraphysiologic serum T levels when administered at the highest FDA-approved dose. Therefore, the investigators' hypothesis is that OT, given at the highest FDA approved dose, will achieve more homogeneous and sustained supraphysiologic levels of serum T that will produce similar or enhanced therapeutic response. To avoid adaptation of CRPC to this sustained level of T, the investigators will utilize a dosing schedule of 1 week-on, 1 week-off.

ELIGIBILITY:
Inclusion Criteria:

* Patient has the ability to understand and willingness to sign a written informed consent document.
* Patient is a male aged 18 years or older.
* Patient has histologically-confirmed adenocarcinoma of the prostate
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2 (as defined in Appendix A: Performance Status Criteria;
* Patient has evidence of metastatic, measurable disease by CT scan. Measurable disease is defined by RECIST 1.1 as at least one measurable lesion ≥10mm by CT scan
* Patient is progressing on continuous androgen ablative therapy (either surgical castration or LHRH agonist/antagonist)
* Patient has documented castrate level of serum testosterone (<50 ng/dl)
* Patient is progressing on luteinizing hormone-releasing hormone (LHRH) agonist/antagonist plus anti-androgen or abiraterone for CSPC. (Note: Must be off anti-androgen or abiraterone for 4 weeks prior to first treatment with OT.) LHRH (luteinizing hormone-releasing hormone)
* Patient has had prior docetaxel for CSPC. Note: Docetaxel is permitted if ≤ 6 doses were given in conjunction with first-line androgen deprivation therapy and >6 months since last dose of docetaxel. (CSPC-castrate sensitive prostate cancer)
* Patient is currently taking prednisone and cannot be weaned entirely off. Note: Patient's dose must be maintained on lowest stable dose that relieves symptoms. Patient is receiving prednisone in conjunction with abiraterone acetate must be weaned off prednisone if possible prior to starting OT.
* Patient has had a rising PSA on two successive measurements at least two weeks apart.
* Patient agrees to continue on castrating therapy throughout OT treatment.
* Patient's screening lab values are within the following parameters:

  1. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 (1.5 ×109/L)
  2. Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
  3. Hemoglobin ≥ 9 g/dL
  4. Serum creatinine < 2.5 times ULN
  5. Bilirubin < 2.5 times institutional upper limit of normal (ULN)
  6. Aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) < 2.5 times ULN
* Patient has had surgery, has completed at least 4 weeks of recovery and has no persistent toxicity > grade 1.

Exclusion Criteria:

* Patient has pain due to metastatic prostate cancer requiring opioid analgesics.
* Patient has had prior treatment with any agent for metastatic castration-resistant prostate cancer. (Includes docetaxel, cabazitaxel, anti-androgen, abiraterone, or investigational agents)
* Patient requires urinary catheterization for voiding due to obstruction secondary to prostatic enlargement thought to be due to prostate cancer or benign prostatic hyperplasia. Note: Patients with indwelling catheter/suprapubic catheter to relieve obstruction are eligible.
* Patient has evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, epidural spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction).
* Patient has evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, epidural spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction).
* Patient has active uncontrolled infection, such as HIV/AIDS or chronic hepatitis B or untreated chronic hepatitis C.
* Patient has had prior history of a thromboembolic event within the past two years and not currently on systemic anticoagulation.
* Patient is on Coumadin. Note: If anticoagulation therapy is mandatory, patient must be switched to an alternative medication) Patients receiving anticoagulation therapy with warfarin, rivaroxaban or apixaban are not eligible for study. [Patients on enoxaparin or edoxaban are eligible for study. Patients on warfarin, rivaroxaban or apixaban, who can be transitioned to enoxaparin prior to starting study treatments, will be eligible.
* Patient has hematocrit >50%, untreated severe obstructive sleep apnea, uncontrolled or poorly controlled heart failure [per Endocrine Society Clinical Practice Guidelines].

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate of Oral Testosterone Undecanoate (CT Scan) | Up to 2 years
  Radiographic responses to Oral Testosterone therapy using CT scan measurements. Radiographic progression is assessed by RECIST (Response Evaluation Criteria in Solid Tumors). Per RECIST, progression is defined as ≥ 20% and ≥ 5 mm from nadir of the sum of the diameters of target lesions.

SECONDARY OUTCOMES:
PSA50 Response to Oral Testosterone Therapy | 2 years
  Number of participants with PSA50 response to Oral Testosterone therapy defined as at least a 50% decline in Prostate Specific Antigen (PSA) from baseline value.
Time to PSA Progression While on Oral Testosterone | Up to 2 years
  Number of weeks from baseline until PSA progression.
Time to Clinical or Radiographic Progression While on Oral Testosterone | Up to 2 years
  Number of weeks from baseline until radiographic or clinical progression, whichever comes first. Radiographic progression is assessed by Response Evaluation Criteria in Solid Tumors (RECIST) and Prostate Cancer Working Group 3 (PCWG3) criteria. Per RECIST, progression is defined as ≥ 20% and ≥ 5 mm from nadir of the sum of the diameters of target lesions. Per PCWG3 criteria, radiographic progression is defined as ≥ 20% sum of the longest diameter of target lesions, or ≥ 2 new lesions on bone scan from baseline. Clinical progression is defined as new spinal cord or nerve root compression, new pathologic fracture or use of opioid analgesics for cancer-related pain.
PSA50 Response to Enzalutamide Therapy | 2 years
  Number of participants with PSA50 response to enzalutamide therapy defined as at least a 50% decline in Prostate Specific Antigen (PSA) from baseline value.
Objective Response Rate of Enzalutamide Therapy (CT Scan) | 2 years
  Radiographic responses to Enzalutamide therapy using CT scan measurements after 3 cycles and after 6 cycles of therapy. Radiographic progression is assessed by RECIST (Response Evaluation Criteria in Solid Tumors) criteria ). Per RECIST, progression is defined as ≥ 20% and ≥ 5 mm from nadir of the sum of the diameters of target lesions.
Peak Testosterone Level | At 4 hours post first dose
  Mean peak testosterone level (ng/dL) measured at 4 hours post first dose of oral testosterone therapy.
Trough Testosterone Level | Up to 96 hours after cycle 1 day 7 dose
  Mean trough testosterone level (ng/dL) measured within 24, 48, 72 or 96 hours after cycle 1 day 7 dose of oral testosterone therapy
PBMC Immunologic and metabolic phenotype | 2 years
  Phenotype of peripheral blood mononucleated cell (PBMC) as defined by number of cluster of differentiation 4 (CD4) Tcells, cluster of differentiation 8 (CD8) Tcells, FOXP3+ Treg cells, B cells, Natural Killer (NK) cells, monocytes, dendritic cells, and myeloid derived suppressor cells. PBMCs will be immunophenotyped using multiparameter flow cytometry.
Change in Quality of Life as Assessed by the-FACIT-Fatigue Questionnaire | 2 years
  The Functional Assessment of Chronic Illness Therapy - Fatigue has a score range of 0-52 with higher scores indicating better quality of life.
Change in Quality of Life as Assessed by the- Short Form 36 (SF-36) Questionnaire | 2 years
  All questions are scored on a scale from 0 to 100. The total score from all of the questions answered is divided by the total number of the questions answered yielding a global score from 0-100 with 100 representing the highest level of functioning possible.
Safety of Trial Therapy as assessed by adverse event reporting | 2 years
  Safety as assessed by adverse event reporting. Grading of adverse events will be done by utilizing the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.03. Determination of relationship of the adverse event to the study procedures or study drug will be performed by the PI using the standard attribution terminology (e.g. unrelated, possibly related, etc.).
Tolerability of Trial Therapy as assessed by adverse event reporting | 2 years
  Tolerability as assessed by adverse event reporting. Grading of adverse events will be done by utilizing the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.03. Determination of relationship of the adverse event to the study procedures or study drug will be performed by the PI using the standard attribution terminology (e.g. unrelated, possibly related, etc.).
Time to PSA Progression While on Enzalutamide | Up to 2 years
  Number of weeks from start of enzalutamide treatment until PSA progression.
Time to PSA Progression While on Enzalutamide from Start of Oral Testosterone Therapy | Up to 2 years
  Number of weeks from start of oral testosterone therapy until PSA progression while on enzalutamide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Allegheny Health Network, Pittsburgh, Pennsylvania